CLINICAL TRIAL: NCT03565250
Title: A Study of Identity Building in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: A Study of Identity Building in Children With ADHD
Acronym: SID-ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Ecole Pratique des Hautes Etudes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-011
Record Dates: First submitted 2018-05-16; First posted 2018-06-21 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Disorder with Hyperactivity; Self concept; Child; Neuropsychology
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADHD patients (Experimental): children aged 8-12 ans with ADHD
  Interventions: Other: self understanding interview
- control (Active Comparator): children aged 8-12 ans without ADHD
  Interventions: Other: self understanding interview

INTERVENTIONS:
Other: self understanding interview — semi-structured interview designed for assessment of identity according to Damon & Hart's 7-dimension develomental model

SUMMARY:
Context: Attention Deficit Hyperactivity Disorder (ADHD), a major public health issue, is a neurodevelopmental disorder characterized by disturbance of attention, pathological impulsivity and a variable level of psychomotor hyperactivity. In addition to medium-term repercussions such as school failure or family dysfunction, these children have difficulties in dealing with emotions, metacognition and self-awareness that have serious consequences for self-regulation and identity construction.

Objective: To investigate identity building in children with ADHD and explore its links with the severity of the disorder and associated neuropsychological disturbances.

Material and method: 20 childrens with ADHD and 20 controls will be recruited over a 24-month period. They will be administered the Damon and Hart's Self-Understanding Interview, exploring 7 identity domains: Physical, Active, Social, Psychological, Continuity, Agentivity, Distinction Self/Other. The severity of ADHD, neuropsychological functioning (attention, working memory, executive functions, long-term memory), self-esteem and internal/external attributive style (locus of control) will be assessed by validated scales. The overall level of identity development and in each dimension will be compared between patients and controls. Within patients, the correlations between level of identity development and the severity of ADHD will be explored, as well as with neuropsychological functioning, with statistical control of age.

Assumptions: The investigators hypothesize that children with ADHD will exhibit a significantly lower level of identity development than controls, which will be positively correlated with neuropsychological functioning, and negatively correlated with the severity of ADHD.

DETAILED DESCRIPTION:
Visit 1: the physician will check inclusion and non-inclusion criteria and co-morbidities of patients and controls using a semi-structured interview (K-SADS-PL). He/She will also assess the overall functioning level of patients and controls (GAF) and will evaluate for patients only the severity of ADHD using ADHD-RS.

Visits number 2 and 3: Cognitive and neuropsychological evaluations:

2 consultations to be distributed in one month depending on the availability of patients (no time limit imposed between the 2 consultations) In order to investigate any cognitive dysfunctions, patients and controls will be referred to the neuropsychologists of the department concerned (pediatrics or child and adolescent psychiatry). They will perform the WISC-V, CPT, Wisconsin SCD, CMS Stories Test. Several questionnaires will be completed by parents and/or children : BRIEF, Self-esteem Questionnaire, Causal Style Questionnaire. This whole assessment will require a total of 2 consultations, one of 1:30 and the second of about 1 hour. Patients on methylphenidate medication should be discontinued the same day during the second session of the neuropsychological check-up.

Visit number 4: Self-Understanding Interview: 1 hour consultation The interview specifically assessing self-understanding will be conducted with children suffering from ADHD and control children. This investigation consists of an interview requiring 1h consultation for which patients should have taken their usual treatment by MPH if necessary. An audio recording of this test will be made.

Inclusion and the first psychological assessment session (visit 1 and visit 2) can be done on the same day. All 3 appointments must be completed in a period of less than 3 months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

Patient group:

* Child aged 8 to 12,
* clinical diagnosis of ADHD according to DSM-V criteria
* Informed consent signed by the holder (s) of the exercise of parental authority and specifying the decision of the child himself,
* Subject having French as mother tongue,
* Subject affiliated to the social security system.

Control group:

* Child aged 8 to 12,
* Not suffering from ADHD according to DSM-V criteria
* Informed consent signed by the holder (s) of the exercise of parental authority and specifying the decision the child himself,
* Subjects with French as their mother tongue,
* Subject affiliated to the social security system.

Exclusion Criteria:

* Sensory disorders,
* Pathology of the brain (head trauma, epilepsy, others),
* Major psychiatric comorbidity (current depressive episode, schizophrenia, bipolar disorder, autism spectrum disorders),
* Anticonvulsant treatment
* Consumption of toxic (drug, alcohol).
* Mental retardation QI less than 70

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2018-07-20 (Estimated); Primary Completion 2020-08-04 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Identity building | baseline
  Self understanding interview (Damon ahd Hart): analysis and developmental characterization of the child's discourse on himself,
  Model distinguishes the two components of Self:
  * the me-self: aggregation of self-knowledge;
  * The I self: the Self-as-subject; the subjective component that performs the act of self-knowledge.
  to attest to identity development:
  * The average level of identity development for me-self as a whole is calculated by summing the total number of segments in each developmental level multiplied by his cardinal, all divided by the total number of segments
  * Breakdown of segments of speech in the 4 modal levels (superficial, self-centered, interactive, codified) for each of the identity dimensions of the component of me-self (Physics, Active, Social, Psychological, Continuity, Agentivity, Distinction Self / Other) ,
  * The best developmental level for each dimension of the I-Self component 0 à 4

SECONDARY OUTCOMES:
• Intensity score of ADHD | baseline
  18 items exploring hyperactivity, impulsivity and inattention symptômes rated on a scale of 4 points:
  * 0: Rarely or never
  * 1: Some times
  * 2: Often
  * 3: Very often
  a score greater than or equal to 28 is required to qualify a significant ADHD. (min=0-max=54)
Self esteem | baseline
  The Child Perception Profile is the French adaptation (Pierrhumbert) of the Self-Perception Profile for Children (Harter).This self-questionnaire for children aged 8 to 13 explores self-esteem through 30 questions about daily life, coded on a scale from 1 to 4. First, the young person chooses the description that looks the most; he then determines how much he looks like him.
  It provides an overall self-esteem score and six sub-scores: academic, social, physical, appearance, driving and self-worth.
  Each dimension is explored by 5 questions, the sub-scores are obtained by adding the items, the overall self-esteem score is obtained by adding the sub-scores.
  The higher the score, the higher the self-esteem
Causal style | baseline
  The Child Causal Style Questionnaire is a self-administered questionnaire that assesses the child's "locus of control", that is, how much does he attribute responsibility for his failures and successes to oneself (internal locus) or to others (external locus). It consists of 24 items describing plausible events, 12 positive and 12 negative, for which the child must choose a cause.
Global Assessment of Functioning Scale | baseline
  The Global Assessment of Functioning (GAF) is a numeric scale used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of an individual, e.g., how well one is meeting various problems-in-living. Scores range from 100 (extremely high functioning) to 1 (severely impaired).
working memory | baseline
  memory of numbers, memory of images in Wechsler Intelligence Scale for Children 5
executive functions | baseline
  BRIEF Wisconsin sorting card test
Long-term memory | baseline
  History recall test (from children memory scale ; Cohen)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Amélie Tordjman-Madigand, MD, Principal Investigator — CHU CAEN
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No